CLINICAL TRIAL: NCT03287687
Title: The Safety and Efficacy of Carbon Dioxide for Insufflation During Endoscopy in Pediatric Patients
Brief Title: Safety and Efficacy of CO2 for Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Warren Bishop (Other)
Responsible Party: Sponsor-Investigator, Warren Bishop, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 201706767
Record Dates: First submitted 2017-09-12; First posted 2017-09-19 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Endoscopy; Insufflation
MeSH Terms: interventions — Carbon Dioxide

STUDY DESIGN:
Intervention Model Description: Double blinded, placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done 1:1, double blinded. - Procedure nurse will randomly choose an envelope from a box; the envelope contains a card listing either "CO2" or "Air". The envelopes will be unmarked and will be prepared with an equal number of cards for each arm. The procedure nurse then turns on either CO2 or air insufflation according to the card in the envelope. The air/CO2 controls will be kept covered to preserve blinding of the endoscopist. She will also record the patient's arm allocation in a logbook, which will be kept in a locked cabinet.
  * These events will precede entry of the patient and endoscopist into the procedure room.
  * Therefore, all study participants are blinded and allocation is also blinded also.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Air for insufflation (Active Comparator): In this arm of patients, air which is currently used as standard of care will be used for insufflation
  Interventions: Drug: Air insufflation
- Carbon dioxide gas for insufflation (Experimental): in this arm of patients, carbon dioxide (CO2) will be used for insufflation during endoscopy
  Interventions: Drug: Carbon dioxide (CO2) gas insufflation

INTERVENTIONS:
Drug: Carbon dioxide (CO2) gas insufflation — CO2 gas use for insufflation during endoscopy instead of air insufflation
  Other Names: CO2
  Arms: Carbon dioxide gas for insufflation
Drug: Air insufflation — Air insufflation is the standard of practice (used in the control arm)
  Other Names: Control
  Arms: Air for insufflation

SUMMARY:
Hypothesis:

Carbon dioxide gas use for endoscopic insufflation is safe and results in less abdominal distension and discomfort; it is equally effective as air in pediatric patients undergoing endoscopic procedures.

Aim 1:

Determine the occurrence and severity of abdominal discomfort and distension associated with endoscopic procedures at baseline, upon awakening from anesthesia, at discharge and at 4 hours after discharge in carbon dioxide group when compared to the air group.

Aim 2:

Determine if the expertise level of the endoscopist contributes to abdominal discomfort and distension following endoscopy, and whether this differs in the carbon dioxide group versus air group.

Aim 3:

Determine if carbon dioxide is as effective as air for insufflation.

DETAILED DESCRIPTION:
STUDY DESIGN: A Prospective, Randomized, Double-Blinded, Controlled Trial We intend to enroll 250 patients aged between 6 months and 21 years in a randomized, double-blind study comparing the use of air (our current routine) vs. carbon dioxide (CO2) for insufflation (inflation) of the gut during endoscopy. The primary endpoint will be abdominal girth and abdominal pain/discomfort after undergoing the endoscopy. Secondary endpoints will be indirect measures of CO2 absorption (respiratory rate and end-tidal CO2)throughout the procedure, determination whether the endoscopist's training level influences the primary endpoint,and determination if CO2 and air are equally effective for adequate intestinal visualization . Similar studies in adults have demonstrated safety and efficacy of CO2 in minimizing bloating and abdominal pain following endoscopy and show no difference in efficacy of insufflation. However, studies done to date in children have not been comprehensive in data gathering and analysis. We now have the capability to routinely use CO2 for insufflation in our new Stead Family Children's Hospital procedure unit, and wish to take this opportunity to fully document both efficacy and safety of CO2 insufflation in children undergoing our most common endoscopic procedures, including esophagogastroduodenoscopy (EGD, upper endoscopy,) colonoscopy, or combined upper endoscopy and colonoscopy. All patients in the study will be sedated by the anesthesia team using propofol as the primary agent. We will exclude patients who are judged to be at risk of respiratory compromise.

Informed consent will be obtained as always for the procedure itself; additional consent and/ assent (when appropriate) will be obtained for study participation. For patients or parents who opt out of the study; air will be used, as per our current routine, for insufflation. Those willing to participate in the study will be randomly assigned to either carbon dioxide or air for insufflation during their endoscopic procedure. Both the endoscopist and patient will be blinded to arm of study.

DATA COLLECTION: At baseline, routine vital signs (HR, BP, RR, oxygen saturation), end tidal CO2, and pain assessment (see below) will be documented. Abdominal girth, measured at the umbilicus, will be documented at baseline as well. The expertise level of the primary endoscopist will be noted; fellow (1st, 2nd, or 3rd year) or faculty will be recorded. A faculty gastroenterologist will be present for the entire procedure.

During the endoscopic procedure, again as per our usual routine, end-tidal CO2 will be continuously monitored and recorded in Epic by the anesthesia team. Other parameters that will be monitored and recorded continuously will include, HR, BP respiratory rate, and oxygen saturation. Based on published studies, we do not anticipate any evidence of detectable CO2 absorption during the procedure, but will be prepared to unblind the study and switch to air insufflation if any concern arises during the procedure. The duration and type of procedure will be noted for all patients.

At the end of the procedure, Heart rate (HR) , Blood pressure (BP), respiratory rate (RR), oxygen saturation, end tidal CO2, abdominal girth, and pain assessment will be documented again. "Breath to breath" analysis of the end tidal CO2 monitor tracing will be performed later, using recorded data, study by Dr. Timothy Starner (Pediatric pulmonologist). This will enable us to determine if there had been any evidence of an increased respiratory rate associated with increased CO2 absorption.

We will use the verbal scale : face, legs, activity, cry, consolability (FLACC) scale to assess pain upon arrival to recovery area. After awakening, abdominal discomfort will be assessed for children who are able to do so, and the assessment will be repeated at discharge from the facility. FLACC will be used for all children with appropriate developmental status, age 5 years and older for normal children. After discharge, the parents will complete an additional brief pain assessment at home at 4 hours after discharge. For those who had an abdominal girth increase of at least 10% from baseline, abdominal girth will be re-measured at home, at 4 hours after discharge.

We will use the non-verbal FLACC scale for children unable to verbally report pain using the visual scale.

Parents will report pain and abdominal girth data done at home by returning a pre-stamped postcard. Those who do not communicate this information will be called by a member of the research team for this information after five working days.

We hypothesize, based on adult and few pediatric studies, that post-procedure abdominal discomfort will be significantly decreased in the CO2 group, and that CO2 will be shown to be safe and effective for endoscopic insufflation.

Efficacy of insufflation will be assessed by the endoscopist immediately after the procedure using a 5-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric gastroenterology patients aged 6 months through 21 years undergoing endoscopic procedures in the Stead Family Children's Hospital (SFCH) Lower Level 2 procedure room or the operating room in the SFCH who willingly consent/ascent to the study. These procedures will range from Esophagogastroduodenoscopy, Colonoscopy, and those having both Esophagogastroduodenoscopy and Colonoscopy.

Exclusion Criteria:

* Non English speaking families who require the services of a translator Children outside the stipulated age range of study. Children in foster care homes or wards of the court. Children and parents who do not willingly consent to the study Children with history of bronchopulmonary dysplasia or other chronic respiratory compromise.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren P Bishop, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Homan M, Mahkovic D, Orel R, Mamula P. Randomized, double-blind trial of CO2 versus air insufflation in children undergoing colonoscopy. Gastrointest Endosc. 2016 May;83(5):993-7. doi: 10.1016/j.gie.2015.08.073. Epub 2015 Sep 10. PMID 26363332
- [Derived] Dike CR, Rahhal R, Bishop WP. Is Carbon Dioxide Insufflation During Endoscopy in Children as Safe and as Effective as We Think? J Pediatr Gastroenterol Nutr. 2020 Aug;71(2):211-215. doi: 10.1097/MPG.0000000000002724. PMID 32304555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 180 procedures were enrolled; 91 procedures in the CO2 group and 89 procedures in the air group.
  There were 178 participants enrolled. 2 participants were enrolled twice
Pre-assignment Details: There were no significant events in this study. There were 178 patients enrolled for 180 procedures. 2 participants were enrolled twice
Units Other Than Participants: Procedures
Groups:
- Air for Insufflation: In this arm of patients, air which is currently used as standard of care will be used for insufflation
  Air: Air is the standard of practice and will be used in the control arm
- Carbon Dioxide Gas for Insufflation: in this arm of patients, carbon dioxide (CO2) will be used for insufflation during endoscopy
  Carbon dioxide gas for insufflation: Carbon dioxide gas use for insufflation during endoscopy instead of air
Period: Overall Study
Arm/Group | Air for Insufflation | Carbon Dioxide Gas for Insufflation
Started | 88; 89 Procedures | 90; 91 Procedures
Procedures | 88; 89 Procedures | 90; 91 Procedures
Completed | 88; 89 Procedures | 90; 91 Procedures
Not Completed | 0; 0 Procedures | 0; 0 Procedures

BASELINE CHARACTERISTICS:
Population: 178 participants enrolled in 180 procedures were blindly randomized to arms air or CO2 insufflation
Groups:
- Total: Total of all reporting groups
Arm/Group | Air for Insufflation | Carbon Dioxide Gas for Insufflation | Total
Number analyzed (Participants) | 88 | 90 | 178
Age, Customized [Number; unit: participants]
  < 4 years | 2 | 6 | 8
  > 4 years | 86 | 84 | 170
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 46 | 99
  Male | 35 | 44 | 79
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 88 | 90 | 178
Weight [Median (Full Range); unit: kilograms] | 47.2 [7.9 to 97.4] | 46.6 [9.4 to 128.5] | 46.9 [7.9 to 128.5]
ASA class status [Number; unit: participants] — Patient's overall health status based on American Society of Anesthesiologists (ASA) classification (ASA class I and II considered low risk sedation population, higher ASA class considered high risk population)
  participants
    Low ASA class (I&II, low sedation risk) | 55 | 65 | 120
    High ASA class (> II high sedation risk) | 33 | 25 | 58
Type of procedure [Number; unit: Participants] — Patients undergoing diagnostic or therapeutic endoscopic procedures were recruited including esophagogastroduodenoscopy only (EGD), combined EGD and colonoscopy, percutaneous endoscopic gastrostomy PEG, and PEG tube exchange. Some participants were included in more than one procedure.
  Participants
    EGD only | 44 | 44 | 88
    EGD/Colonoscopy | 30 | 30 | 60
    Any Colonoscopy | 36 | 33 | 69
    Other | 9 | 14 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Abdominal Distension
Description: Change in abdominal girth from baseline to end of procedure (Time Difference 1) or Change in abdominal girth from baseline to time of discharge ((Time Difference 2)
Time Frame: Mean change in abdominal girth between time points were compared between groups
Population: 178 participants were enrolled for 180 procedures
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Procedures
Arm/Group | Air for Insufflation | Carbon Dioxide Gas for Insufflation
Number analyzed (Participants) | 88 | 90
Number analyzed (Procedures) | 89 | 91
cm
  Time Difference 1: Difference from baseline to end of procedure (median 16 minutes), cm | 0.9 (2.3) | 0.5 (2.0)
  Time Difference 2: Difference from baseline to discharge (approximately 120 minutes), cm: number analyzed (Participants) | 60 | 60
  Time Difference 2: Difference from baseline to discharge (approximately 120 minutes), cm | 1.1 (2.2) | 0.9 (2.5)

2. Secondary Outcome: Elevations of End Tidal Carbon Dioxide
Description: Number of Procedures with Elevated End Tidal CO2 level (≥ 60 mmHg)
Time Frame: Time frame of monitoring from start to end of procedure (average of 12 minutes for EGD procedures)
Population: 178 participants were included in 180 procedures
Measure: Number; unit: Procedures
Units Other Than Participants: Procedures
Arm/Group | Air for Insufflation | Carbon Dioxide Gas for Insufflation
Number analyzed (Participants) | 88 | 90
Number analyzed (Procedures) | 89 | 91
Procedures | 5 | 34

3. Secondary Outcome: Procedures With Post Endoscopy Reported Symptoms
Description: Procedures with post endoscopy reported symptoms, up to 4 hours, of belching, bloating and flatulence
Time Frame: Frequency of reported symptoms up to 4 hours post endoscopy was compared between groups
Population: 178 participants were enrolled for 180 procedures
Measure: Number; unit: procedures
Units Other Than Participants: Procedures
Arm/Group | Air for Insufflation | Carbon Dioxide Gas for Insufflation
Number analyzed (Participants) | 88 | 90
Number analyzed (Procedures) | 89 | 91
procedures
  Belching: number analyzed (Procedures) | 60 | 60
  Belching | 18 | 31
  Bloating: number analyzed (Procedures) | 60 | 60
  Bloating | 13 | 5
  Flatulence: number analyzed (Procedures) | 60 | 60
  Flatulence | 26 | 9

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from start of procedure time up to 4 hours post procedure
Description: All cause Mortality Procedural related adverse events included bleeding and perforation Anesthesia related adverse events reported included hypoxia and aspiration
Arm/Group | Air for Insufflation | Carbon Dioxide Gas for Insufflation
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/90
Other Adverse Events (participants affected / at risk) | 1/88 | 4/90
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Air for Insufflation (N=88) | Carbon Dioxide Gas for Insufflation (N=90)
Procedural related complication - Bleeding (Gastrointestinal disorders) | 0 (0) | 2 (2) — Bleeding
Anesthesia related complication - Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Aspiration
Anesthesia related complication - Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Hypoxia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03287687/Prot_002.pdf
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03287687/SAP_003.pdf